CLINICAL TRIAL: NCT04385407
Title: Sofosbuvir in Combination With Ribavirin or Simeprevir: Real-life Study of Patients With Hepatitis C Genotype 4
Brief Title: Sofosbuvir With Ribavirin or Simeprevir With HCV GT4 Egyptian Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOF-SMV-RBV
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Egyptian patients; HCV GT4; Naive; Ribavirin; Simeprevir; Sofosbuvir; Experinced
MeSH Terms: interventions — Sofosbuvir; Simeprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SOF + RBV (Naive) (Active Comparator): For treatment-naive participants, SOF was given in a dose of 400 mg/day + RBV was given orally in the morning and in the evening (total daily dose was based on body weight:<75 kg, 1000 mg; >75 kg, 1200 mg).
  Interventions: Drug: Sofosbuvir + Simeprevir + Ribavirin
- SOF + RBV (Experienced) (Active Comparator): For treatment-experienced participants, SOF was given in a dose of 400 mg/day + RBV was given orally in the morning and in the evening (total daily dose was based on body weight:<75 kg, 1000 mg; >75 kg, 1200 mg).
  Interventions: Drug: Sofosbuvir + Simeprevir + Ribavirin
- SOF + SMV (Naive) (Active Comparator): For treatment-naive participants, SOF was given in a dose of 400 mg/day + SMV orally as a single 150 mg q.d. capsule.
  Interventions: Drug: Sofosbuvir + Simeprevir + Ribavirin
- SOF + SMV (Expereined) (Active Comparator): For treatment-experienced participants, SOF was given in a dose of 400 mg/day + SMV orally as a single 150 mg q.d. capsule.
  Interventions: Drug: Sofosbuvir + Simeprevir + Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir + Simeprevir + Ribavirin
  Other Names: Olysio is a trade name of simeprevir; Sovaldi is a trade name of sofosbuvir

SUMMARY:
A total of 201 participants with chronic HCV GT4 infection were allocated into two groups. One group participants were treated with SOF plus RBV (24 weeks). The second group was treated with SOF plus SMV (12 weeks).

DETAILED DESCRIPTION:
A total of 201 participants, treatment-naïve and experienced, with chronic HCV GT4 infection were allocated into two groups based on the type of the regimen used. All eligible participants were treated orally with SOF plus daily oral weight-based RBV (24 weeks; group 1), or SOF plus daily oral SMV (12 weeks; group 2).

ELIGIBILITY:
Inclusion Criteria:

* Participants with plasma HCV RNA level >10,000 IU/L for the two groups.
* Treatment-experienced patients in group 1 were those who had previously failed treatment with classical peg-IFN/RBV therapy.
* Treatment-experienced patients in group 2 were those who had previously failed treatment with SOF/RBV

Exclusion Criteria:

* coinfected with hepatitis B virus or human immunodeficiency virus infection,
* any cause of liver disease other than HCV GT4 infection;
* liver decompensation,
* hepatocellular carcinoma,
* major severe illness, such as renal failure, congestive heart failure, thyroid dysfunction, respiratory failure, autoimmune disease and poorly controlled diabetes (HbA1C >9)
* Participants with blood picture abnormalities, such as anemia (hemoglobin concentration of 10 g/or less) and thrombocytopenia (platelet count <50,000 cells/mm3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With HCV 12 | 12 weeks after last dose
  HCV 12 is HCV RNA level <15 IU/mL at 12 weeks after planned end of treatment (EOT).
Number of Participants With Adverse Events | up for 12 weeks after planned EOT.
  An adverse event (AE) is defined as any untoward medical occurrence in a participant clinical investigation administered the drugs of the study.
  A serious adverse event (SAE) is an event that results in death, life-threatening, participant hospitalization, or disability/incapacity

SECONDARY OUTCOMES:
Percentage of Participants With Virologic relapse | 12 weeks after the last dose
  Viral relapse was HCV RNA level <15 IU/mL at EOT, but >15 IU/mL levels through 12 weeks after planned EOT
Percentage of Participants With Virologic null response | 24 or 36 weeks stating from the first dose
  Virologic null response is defined as HCV RNA >15 IU/mL levels throughout the entire treatment period

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Moneim A, Aboud A, Abdel-Gabbar M, Zanaty MI, Elbary AAA, Ramadan M. Sofosbuvir in combination with ribavirin or simeprevir: real-life study of patients with hepatitis C genotype 4. Ann Gastroenterol. 2019 Jan-Feb;32(1):93-98. doi: 10.20524/aog.2018.0327. Epub 2018 Nov 24. PMID 30598598
- See also: This link describes the effectiveness and safety of two regimens sofosbuvir (SOF) in combination with either ribavirin (RBV) or simeprevir (SMV) in chronic hepatitis C (CHC) genotype (GT) 4 patients in Egypt. — http://www.annalsgastro.gr/files/journals/1/earlyview/2018/ev-11-2018-08-AG4308-0327.pdf